CLINICAL TRIAL: NCT03736356
Title: Prospective Evaluation of Health Outcomes in AE Casualties: a Pilot Study
Brief Title: Long-term Health Outcomes of AE Casualties
Status: Terminated | Type: Observational
Why Stopped: The study was terminated due to the current COVID-19 pandemic.
Sponsor: Ian Stewart (U.S. Federal Agency)
Collaborators: Naval Health Research Center (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Ian Stewart, Chief, Combat Nephrology, David Grant U.S. Air Force Medical Center
Organization: David Grant U.S. Air Force Medical Center (U.S. Federal Agency)
Other Study IDs: FWH20200146H
Record Dates: First submitted 2018-10-23; First posted 2018-11-09 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Long Term Adverse Effects; Combat Disorders
Keywords: Aeromedical Evacuation; Combat Injury
MeSH Terms: conditions — Long Term Adverse Effects; Combat Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: None Retained — Urine and blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study involves individuals who are currently participating in the Wounded Warrior Recovery Project and underwent aeromedical evacuation (AE) due to injury during deployment in Iraq or Afghanistan. The goal of the study is to understand how best to engage wounded warriors in research activities studying long-term health. Based on the results from this study, the investigators can plan a larger study with the goal to better understand the long-term health conditions of individuals who were injured in combat and improve patient care.

As part of the study, participants will be asked to provide two sets of lab work over the course of a year. Each set of lab work will include one blood draw, one urine sample, and height, weight, and blood pressure measurements. In order to track long-term health, information from participants' lab work will be linked with study-related health data, as well as surveys they have completed with the Wounded Warrior Recovery Project (WWRP).

ELIGIBILITY:
Inclusion Criteria:

1. Combat injury during or after October 2001
2. Aged > 18 years
3. Listed in EMED
4. Underwent AE
5. Enrolled in Wounded Warrior Recovery Project

Exclusion Criteria:

1. Non-battle injury
2. Not listed in EMED
3. Combat injury before October 2001
4. Did not undergo AE
5. Not enrolled in Wounded Warrior Recovery Project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be enrolled in the Wounded Warrior Recovery Project and have a record of aeromedical evacuation (AE) due to combat injury in the Expeditionary Medical Encounter database (EMED). Only those who were injured in combat during or after October 2001 and who are currently >18 years old will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Number of enrolled participants who complete both sets of lab work | Approximately one year from beginning of study participation
  Whether or not enrolled participants complete labs as requested at year 1 and year 2

SECONDARY OUTCOMES:
Complete blood count (CBC) | Approximately one year from beginning of study participation
  Results from this lab test will be used to define physical health outcomes of patients who have transited through the aeromedical evacuation system.
Comprehensive metabolic panel | Approximately one year from beginning of study participation
  Results from this lab test will be used to define physical health outcomes of patients who have transited through the aeromedical evacuation system.
Hemoglobin A1c | Approximately one year from beginning of study participation
  Results from this lab test will be used to define physical health outcomes of patients who have transited through the aeromedical evacuation system.
Cystatin C | Approximately one year from beginning of study participation
  Results from this lab test will be used to define physical health outcomes of patients who have transited through the aeromedical evacuation system.
High sensitivity C-reactive protein (hs-CRP) | Approximately one year from beginning of study participation
  Results from this lab test will be used to define physical health outcomes of patients who have transited through the aeromedical evacuation system.
B Type Natriuretic Peptide (BNP) | Approximately one year from beginning of study participation
  Results from this lab test will be used to define physical health outcomes of patients who have transited through the aeromedical evacuation system.
Urine microalbumin/creatinine ratio | Approximately one year from beginning of study participation
  Microalbumin and creatinine will be combined obtain this ratio in mcg/mg creatinine. Results from this lab test will be used to define physical health outcomes of patients who have transited through the aeromedical evacuation system.
Blood pressure | Approximately one year from beginning of study participation
  Blood pressure measurements will be used to define physical health outcomes of patients who have transited through the aeromedical evacuation system.
Responses from Wounded Warrior Recovery Project surveys | Approximately one year from beginning of study participation
  Surveys included in this study will include the most recent Wounded Warrior Recovery Project survey prior to study enrollment, the six month followup survey, and the one year followup survey.
Height | Approximately one year from beginning of study participation
  Height in feet. This measurement will be used to define physical health outcomes of patients who have transited through the aeromedical evacuation system.
Weight | Approximately one year from beginning of study participation
  Weight in pounds. This measurement will be used to define physical health outcomes of patients who have transited through the aeromedical evacuation system.

CONTACTS AND LOCATIONS:
Overall Officials: Ian J Stewart, MD, Principal Investigator — David Grant USAF Medical Center
Locations (1):
- David Grant USAF Medical Center, Travis Air Force Base, California, United States

IPD SHARING:
Plan to Share IPD: No